CLINICAL TRIAL: NCT04674202
Title: Pilot Study: Comparison of Patients' Knowledge of Direct Oral Anticoagulants in Post-hospitalization Between 2 Cardiology Departments Offering or Not a Pharmaceutical Interview During Hospitalization
Acronym: EDUC-AOD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PPRC08; 2020-A02285-34 (Other: IDRCB)
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Direct oral anticoagulants
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pharmaceutical interview: This group will benefit from a pharmaceutical interview, accordingly with the common practice in the department in which they are treated.
  Interventions: Other: Phone interview
- No pharmaceutical interview: This group will not benefit from a pharmaceutical interview, accordingly with the common practice in the department in which they are treated.
  Interventions: Other: Phone interview

INTERVENTIONS:
Other: Phone interview — The participant will have 2 phone interview in which they will be asked about their knowledge of direct oral anticoagulants.

SUMMARY:
Direct oral anticoagulants (Rivaroxaban, Apixaban and Dabigatran) are an alternative to anti-vitamin K drugs and low molecular weight heparins in many cardiovascular diseases.

This new class of anticoagulants represents a particular and very promising advance: they are administered orally, their mechanism of action is rapid and direct on coagulation and their predictable pharmacological action allows for administration at fixed doses. In contrast to anti-vitamin K, there is no need for routine biological monitoring.

However, their therapeutic range is narrow and there is no routine biological monitoring. Rigorous compliance is therefore necessary. In addition, there are no official validated recommendations either for the measurement of anticoagulant activity in certain emergency situations, or for the management of severe bleeding (except recently for Pradaxa®).

Their correct use requires the training and involvement of health professionals as well as information and support for patients.

Pharmaceutical interviews are one of the main ways in which pharmacists can ensure this security through personalized and optimal patient care.

The purpose of these interviews is to:

* Reinforce the pharmacist's advisory, educational and preventive roles with patients;
* To enhance the pharmacist's expertise in the area of medication;
* To evaluate the patient's knowledge of his or her treatment;
* To assess the patient's knowledge of his or her treatment; To seek the patient's therapeutic adherence and help him or her to take ownership of his or her treatment;
* To evaluate, in the long term, the patient's appropriation of his or her treatment.

In this way, they enable involvement with patients while providing a link between healthcare professionals, which is essential for optimal patient care.

In recent years, numerous studies have been conducted on pharmaceutical interviews in the United Kingdom and the Netherlands.

On the other hand, few studies have been conducted in France to evaluate the clinical impact of pharmaceutical interviewing in medical services.

The aim of this study is to compare patients' knowledge of direct oral anticoagulants between 2 cardiology departments offering or not a pharmaceutical interview.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for more than 48 hours in a cardiology department with a discharge prescription for curative anticoagulation.
* Indication for a direct oral anticoagulant for atrial fibrillation, deep vein thrombosis or pulmonary embolism

Exclusion Criteria:

* Patients treated for the prevention of venous thromboembolic disease who have undergone scheduled total hip replacement or total knee replacement surgery.
* Patient with cognitive impairment
* Patients with a previous prescription for a direct oral anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of patients hospitalized in a cardiology department with a discharge prescription for direct oral anticoagulants.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a "satisfactory" knowledge score 3 months after hospital discharge | 3 months after hospital discharge
  Knowledge of direct oral anticoagulants will be assessed with a 4 item questionnaire. The score ranges from 0 "no knowledge" to ≥ 3 "satisfactory knowledge".

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal de Montreuil, Montreuil
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé

IPD SHARING:
Plan to Share IPD: Undecided